CLINICAL TRIAL: NCT04373798
Title: Triage Strategies Based on C-reactive Protein Levels Among Individuals With COVID-19: A Prospective Cohort Study
Brief Title: C-reactive Protein Levels Among Individuals With COVID-19
Status: Completed | Type: Observational
Sponsor: Henning Bliddal (Other)
Responsible Party: Sponsor-Investigator, Henning Bliddal, Professor, Frederiksberg University Hospital
Organization: Frederiksberg University Hospital (Other)
Other Study IDs: APPI2-CV-2020-02
Record Dates: First submitted 2020-05-01; First posted 2020-05-04 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Coronavirus Infection
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspected COVID-19: Individuals with symptoms who are seen at covid19 check points for covid19 diagnosis.
  Interventions: Diagnostic Test: C-reactive protein

INTERVENTIONS:
Diagnostic Test: C-reactive protein — Measurement of CRP value from blood sample taken at covid19 check point (baseline).

SUMMARY:
The primary objective of this multi-center study is to clarify the value of a CRP measurement for triage of patients initially presenting with light symptoms of the COVID-19 infection.

Current recommendations of management of COVID-19 include large-scale tests for virus. Such tests reveal whether an individual is infected with the virus, however, the demonstration of virus per se has no prognostic value for the ensuing course of the COVID-19 disease. Publications of possible treatments strategies increase exponentially, while evidence of triage of the affected individuals is mainly based on the level of pulmonary affection as measured by the Oxygen saturation.

To inform decision making for which patients are to be hospitalized due to risk of developing more severe affection, this study addresses the question, whether triage may be performed with the aid of a simple CRP measurement.

ELIGIBILITY:
Inclusion Criteria:

1. A test for COVID-19 taken at the check point
2. Signed, informed consent for blood test to be drawn for the Biobank

Exclusion Criteria:

1. Former admission to hospital for COVID-19
2. Direct admission from check point.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who are COVID-19 positive at the check point test.
Sampling Method: Non-Probability Sample
Enrollment: 1006 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Hospitalisation | within 28 days
  Admission to a hospital. Reason for admission is recorded.

SECONDARY OUTCOMES:
Death | within 28 days
Transfer to Intensive Care Unit | within 28 days
Oxygen treatment during hospitalisation | within 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Henning Bliddal, DMSc, Principal Investigator — The Parker Institute
Locations (1):
- The Parker Institute, Frederiksberg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided